CLINICAL TRIAL: NCT06502249
Title: Modulatory Effect of Prodigiosin or Pioglitazone on Tumor Immune Microenvironment and the Crosstalk to Immune-Checkpoint Protein(s)
Brief Title: Modulatory Effect of Prodigiosin or Pioglitazone on TIME and the Crosstalk to Immune-Checkpoint Protein(s)
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Prof. Nadia M. Hamdy, Ph.D., Professor of biochemistry and molecular biology, Ain Shams University
Other Study IDs: P#2
Record Dates: First submitted 2024-06-12; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer; NSCLC
Keywords: Immune checkpoint proteins; pioglitazone; prodigiosin; TIME
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected and stored at -20°c. RNA will then be extracted followed by cDNA synthesis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: Healthy volunteers not suffering from any disease or not taking any Medications
- Diseased: NSCLC patients

SUMMARY:
Lung cancer is one of the most common and serious types of cancer. Lung tumor cells exploit immune checkpoint proteins (ICPs) to maintain immune tolerance and thus promote tumor progression and invasion. Inhibition of ICPs using antibody therapies is one of the most common approaches for the treatment of lung cancer. Unfortunately, these antibody-based therapies can lead to severe adverse events. Moreover, a significant number of patients do not respond to immune checkpoint inhibition due to tumor heterogeneity and the immunosuppressive tumor immune microenvironment (TIME). The use of small molecule targeted approach instead of antagonizing antibodies may have the potential advantage of being able to target multiple ICPs in TIME with a single agent as well as improved tumor distribution.

DETAILED DESCRIPTION:
1. Introduction 1.1. Background Components of the tumor microenvironment (TME) presented by immune cells, tumor cells, and their derived factors are known as Tumor immune microenvironment (TIME). Tumors can gradually shape TIME into an immunosuppressive state to hinder host immunity. Two opposing immune responses help shape TIME. One side of the immune cells represented by M1 macrophage, T-lymphocyte, Dendritic cells (DC), and Natural killer cells (NK) play a role in the antitumor immune response. On the contrary, tumor-promoting immune cells represented by regulatory T cells (Treg), myeloid-derived suppressor cells (MDSC), M2 macrophage, and group 2 innate lymphoid cells (ILC2) contribute to an immunosuppressive microenvironment.

Under physiological conditions, several immune checkpoint proteins (ICPs) are expressed on various immune cells. These ICPs bind to their complementary ligand to activate T-cells' inhibitory signals, therefore they act as gatekeepers for normal cells. Among the first immune checkpoint proteins discovered were cytotoxic T-lymphocyte antigen number 4 (CTLA-4) and programmed cell death protein 1 (PD-1).. Recently, several immune checkpoint proteins have been discovered; T-cell immunoglobulin domain and mucin domain-containing molecule-3 (TIM-3), T-cell immunoglobulin and ITIM domain (TIGIT), B and T cell lymphocyte attenuator (BTLA), lymphocyte activation gene (LAG3) and V-domain Ig suppressor of T cell activation (VISTA). Unfortunately, tumor and tumor-promoting immune cells exploit these ICPs to escape immune system-mediated cell death.

Several factors could control the expression of ICPs. HSP90 chaperone function plays a role in the regulation of immune cell function by controlling ICPs expression. Zavareh and his colleagues showed that HSP90 inhibitors have a direct inhibitory effect on the expression of ICPs including PD-L1 and PD-L2. Only one study implicated prodigiosin inhibitory effect on HSP90, yet, the effect of prodigiosin on novel immune checkpoint proteins and its modulatory effect on TIME via HSP90 has not been investigated.

The expression of ICPs has also been shown to be controlled by the IL-6/JAK2/STAT3 pathway. High levels of STAT3 and JAK2 levels have been attributed to poor prognosis in non-small cell lung cancer (NSCLC) patients. c-MYC, one of the downstream targets of IL-6/STAT3 signaling, could promote tumor immune escape by increasing the levels ICPs . Pioglitazone, a peroxisome proliferator-activated receptor-γ agonist, inhibited c-MYC-mediated immune escape by inducing PD-L1 protein degradation. Pioglitazone could enhance cancer immunotherapy and T-cell activation by decreasing PD-L1 protein levels . The inhibitory effect of pioglitazone on STAT3 has been studied in different types of cancer . However, the modulatory effect of pioglitazone on novel ICPs via the IL-6/STAT3 pathway and c-MYC remains to be investigated.

1.2. PROBLEM. 1.2.1.Lung Cancer is the leading cause of cancer death in both men and women aged 50 years and older. The response rate to current ICIs used for the treatment of lung cancer is far from satisfactory.

1.2.2. Cancer cells escape from immune surveillance through "immune-editing". Further research is needed for a better understanding of different immune aspects of lung cancer, including immune escape, immunosuppression, immune editing, and tumor-intrinsic adaptive response.

3. Proposal state of the art: 3.1. TIME is a dynamic process and despite heterogeneity across different cancer types and populations, the role of TIME in tumor progression is similar. 3.2. The expression of ICPs could be regulated by HSP90, IL-6/JAK2/STAT3 Pathway, and c-MYC. Thus, HSP90 inhibition by prodigiosin as well as IL-6/STAT3 and c-MYC inhibition by pioglitazone could have the potential to enhance immune surveillance and immune checkpoint protein blockade therapy.

4. Aim of the work: 4.1. Measuring gene and protein expression of Heat shock Protein 90 (HSP90), IL-6, STAT3, c-MYC and novel immune checkpoint proteins from non-small cell lung cancer (NSCLC) patients.

4.2. Studying the effect of prodigiosin on HSP90and pioglitazone of IL-6/STAT3 and c-MYC for modulating TIME via the expression of one of the novel immune checkpoint proteins.

4.3. Investigate the difference in expression at both protein and mRNA levels following treatment of prodigiosin and pioglitazone on lung cancer cell line(s) (A549 or H460 or Calu-3).

4.4. Loading both drugs in nano-sized particles (NPs) and testing the efficacy against lung cancer cell model both in-vivo and in-vitro.

5. Research objectives: 5.1. Main objectives:

Identifying and targeting promising molecular targets to help eradicate lung tumor cells and prevent the development of treatment resistance or immune resistance.

5.2. Secondary objectives:

5.2.1. Studying the cytotoxic effect of prodigiosin and pioglitazone on lung cancer cell line and in vitro safety assay towards normal human retina pigmented epithelial (RPE1) cell line.

5.2.2. Identification of cell surface markers expressed by various immune cells on lung cancer cell lines (A549 or H460 or Calu-3) using flow cytometry.

5.2.3. Cell treatment with prodigiosin and HSP90 transfection in lung cancer cell lines for further investigation of the modulatory effect of Prodigiosin on TIME.

5.2.4. Cell treatment with pioglitazone and c-MYC transfection or using JAK2/STAT3 inhibitor in lung cancer cell lines for further investigation of the modulatory effect of Pioglitazone on TIME.

5.2.5. Gene expression and measuring protein levels of HSP90 and the novel immune checkpoint proteins before and after the addition of prodigiosin in lung cancer cell line.

5.2.6. Gene expression and measuring protein levels of IL-6, STAT3, c-MYC, and the novel immune checkpoint proteins before and after the addition of pioglitazone in lung cancer cell line.

5.2.7. Studying the in-vivo and in-vitro effects of drug-load nanoparticles in lung cancer model.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 50 years old with NSCLC.

Exclusion Criteria:

* Lung cancer patients with any cancer other than NSCLC
* Lung cancer patients with incomplete data or incomplete histopathology diagnosis report.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Lung cancer patients diagnosed with non-small cell lung cancer and healthy volunteers not suffering from any disease will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Gene Expression (mRNA levels) | 36 months
  mRNA levels of HSP90, IL-6, STAT3,c-MYC and the novel immune checkpoint proteins by qRT-PCR from blood samples collected from NSCLC patients and cell pellets collected from lung cancer cell lines before and after pioglitazone or prodigiosin treatment
Gene Expression (Protein levels) | 36 months
  Protein levels of HSP90, IL-6, STAT3,c-MYC and the novel immune checkpoint proteins by immunoblotting from blood samples collected from NSCLC patients and cell pellets collected from lung cancer cell lines before and after pioglitazone or prodigiosin treatment
cytotoxic effect | 36 months
  Cytotoxic effect of prodigiosin or pioglitazone on lung cancer cell line using MTT assay
Anti-cancer efficiency of drug-loaded nanoparticles | 36 months
  Anticancer efficiency against lung cancer in vivo model using Urethan as lung cancer inducer or in vitro lung cancer cell line

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Hamdy, PhD, Principal Investigator — Faculty of pharmacy Ain Shams university
Locations (1):
- Faculty of Pharmacy, Ain Shams University, Advanced Biochemistry Research Lab, Cairo, Egypt

REFERENCES:
- [Background] Abdelhamed S, Ogura K, Yokoyama S, Saiki I, Hayakawa Y. AKT-STAT3 Pathway as a Downstream Target of EGFR Signaling to Regulate PD-L1 Expression on NSCLC cells. J Cancer. 2016 Jul 18;7(12):1579-1586. doi: 10.7150/jca.14713. eCollection 2016. PMID 27698894
- [Background] Anwar MM, Shalaby M, Embaby AM, Saeed H, Agwa MM, Hussein A. Prodigiosin/PU-H71 as a novel potential combined therapy for triple negative breast cancer (TNBC): preclinical insights. Sci Rep. 2020 Sep 7;10(1):14706. doi: 10.1038/s41598-020-71157-w. PMID 32895397
- [Background] Casey SC, Baylot V, Felsher DW. MYC: Master Regulator of Immune Privilege. Trends Immunol. 2017 Apr;38(4):298-305. doi: 10.1016/j.it.2017.01.002. Epub 2017 Feb 21. PMID 28233639
- [Background] Fu S, Liu Y, Zhang Z, Mei M, Chen Q, Wang S, Yang X, Sun T, Ma M, Xie W. Identification of a Novel Myc-Regulated Gene Signature for Patients with Kidney Renal Clear Cell Carcinoma. J Oncol. 2022 Dec 26;2022:3487859. doi: 10.1155/2022/3487859. eCollection 2022. PMID 37342680
- [Background] Gao FY, Li XT, Xu K, Wang RT, Guan XX. c-MYC mediates the crosstalk between breast cancer cells and tumor microenvironment. Cell Commun Signal. 2023 Jan 31;21(1):28. doi: 10.1186/s12964-023-01043-1. PMID 36721232
- [Background] Gou Q, Che S, Chen M, Chen H, Shi J, Hou Y. PPARgamma inhibited tumor immune escape by inducing PD-L1 autophagic degradation. Cancer Sci. 2023 Jul;114(7):2871-2881. doi: 10.1111/cas.15818. Epub 2023 Apr 24. PMID 37096255
- [Background] Harada D, Takigawa N, Kiura K. The Role of STAT3 in Non-Small Cell Lung Cancer. Cancers (Basel). 2014 Mar 26;6(2):708-22. doi: 10.3390/cancers6020708. PMID 24675568
- [Background] Jia X, Qian J, Chen H, Liu Q, Hussain S, Jin J, Shi J, Hou Y. PPARgamma agonist pioglitazone enhances colorectal cancer immunotherapy by inducing PD-L1 autophagic degradation. Eur J Pharmacol. 2023 Jul 5;950:175749. doi: 10.1016/j.ejphar.2023.175749. Epub 2023 Apr 25. PMID 37105516
- [Background] Lv B, Wang Y, Ma D, Cheng W, Liu J, Yong T, Chen H, Wang C. Immunotherapy: Reshape the Tumor Immune Microenvironment. Front Immunol. 2022 Jul 6;13:844142. doi: 10.3389/fimmu.2022.844142. eCollection 2022. PMID 35874717
- [Background] Mbofung RM, McKenzie JA, Malu S, Zhang M, Peng W, Liu C, Kuiatse I, Tieu T, Williams L, Devi S, Ashkin E, Xu C, Huang L, Zhang M, Talukder AH, Tripathi SC, Khong H, Satani N, Muller FL, Roszik J, Heffernan T, Allison JP, Lizee G, Hanash SM, Proia D, Amaria R, Davis RE, Hwu P. HSP90 inhibition enhances cancer immunotherapy by upregulating interferon response genes. Nat Commun. 2017 Sep 6;8(1):451. doi: 10.1038/s41467-017-00449-z. PMID 28878208
- [Background] Proia DA, Kaufmann GF. Targeting Heat-Shock Protein 90 (HSP90) as a Complementary Strategy to Immune Checkpoint Blockade for Cancer Therapy. Cancer Immunol Res. 2015 Jun;3(6):583-9. doi: 10.1158/2326-6066.CIR-15-0057. Epub 2015 May 6. PMID 25948551
- [Background] Qin S, Xu L, Yi M, Yu S, Wu K, Luo S. Novel immune checkpoint targets: moving beyond PD-1 and CTLA-4. Mol Cancer. 2019 Nov 6;18(1):155. doi: 10.1186/s12943-019-1091-2. PMID 31690319
- [Background] Rahmy S, Mishra SJ, Murphy S, Blagg BSJ, Lu X. Hsp90beta inhibition upregulates interferon response and enhances immune checkpoint blockade therapy in murine tumors. Front Immunol. 2022 Oct 20;13:1005045. doi: 10.3389/fimmu.2022.1005045. eCollection 2022. PMID 36341371
- [Background] Rebe C, Ghiringhelli F. STAT3, a Master Regulator of Anti-Tumor Immune Response. Cancers (Basel). 2019 Aug 30;11(9):1280. doi: 10.3390/cancers11091280. PMID 31480382
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Tokhanbigli S, Alavifard H, Asadzadeh Aghdaei H, Zali MR, Baghaei K. Combination of pioglitazone and dendritic cell to optimize efficacy of immune cell therapy in CT26 tumor models. Bioimpacts. 2023;13(4):333-346. doi: 10.34172/bi.2022.24209. Epub 2022 Aug 9. PMID 37645031
- [Background] Tsubaki M, Takeda T, Tomonari Y, Kawashima K, Itoh T, Imano M, Satou T, Nishida S. Pioglitazone inhibits cancer cell growth through STAT3 inhibition and enhanced AIF expression via a PPARgamma-independent pathway. J Cell Physiol. 2018 Apr;233(4):3638-3647. doi: 10.1002/jcp.26225. Epub 2017 Nov 10. PMID 29030979
- [Background] Xu L, Che S, Chen H, Liu Q, Shi J, Jin J, Hou Y. PPARgamma agonist inhibits c-Myc-mediated colorectal cancer tumor immune escape. J Cell Biochem. 2023 Aug;124(8):1145-1154. doi: 10.1002/jcb.30437. Epub 2023 Jul 2. PMID 37393598
- [Background] Zavareh RB, Spangenberg SH, Woods A, Martinez-Pena F, Lairson LL. HSP90 Inhibition Enhances Cancer Immunotherapy by Modulating the Surface Expression of Multiple Immune Checkpoint Proteins. Cell Chem Biol. 2021 Feb 18;28(2):158-168.e5. doi: 10.1016/j.chembiol.2020.10.005. Epub 2020 Oct 27. PMID 33113406
- [Background] Zhang N, Zeng Y, Du W, Zhu J, Shen D, Liu Z, Huang JA. The EGFR pathway is involved in the regulation of PD-L1 expression via the IL-6/JAK/STAT3 signaling pathway in EGFR-mutated non-small cell lung cancer. Int J Oncol. 2016 Oct;49(4):1360-8. doi: 10.3892/ijo.2016.3632. Epub 2016 Jul 26. PMID 27499357